CLINICAL TRIAL: NCT03492411
Title: Evaluating an eHealth Breastfeeding Resource for Mothers, Fathers, Partners and Co-parents
Brief Title: Evaluating an eHealth Breastfeeding Resource
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ontario Institute of Technology (Other)
Collaborators: Durham Region Health Department (Other)
Responsible Party: Principal Investigator, Jennifer Abbass-Dick, Assistant Professor, University of Ontario Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: v3vt62d9
Record Dates: First submitted 2018-02-22; First posted 2018-04-10 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Breastfeeding, Exclusive; Breastfeeding
Keywords: Breastfeeding; Co-parenting; eHealth; patient education; fathers
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: 150 couples will be randomized to group allocation, intervention group or control group with use sequentially numbered opaque envelopes
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to group allocation. Follow up data will be collected via online survey or telephone interview with survey questions. Mode of data collection will depend on participant preference
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth Intervention (Experimental): This group will receive information about an eHealth breastfeeding co-parenting resource. They will have a short demonstration of the site and will receive weekly emails for 6 weeks reminding them about the resource and their participation in the study.
  Interventions: Other: eHealth Breastfeeding Co-parenting Resource
- Usual Care (No Intervention): This group will not receive any intervention. They will receive emails for 6 weeks reminding them that they are in the study.

INTERVENTIONS:
Other: eHealth Breastfeeding Co-parenting Resource — The eHealth breastfeeding co-parenting resource was designed using a participatory model in partnership with the target population. It contains extensive information about breastfeeding and co-parenting. The topics include not only the importance of breastfeeding and technique but also information on how to manage common issues during breastfeeding establishment as well as over the child's first years, since breastfeeding is recommended to two years and beyond. Interactive learning elements, videos, and links to additional resources are included in the resources.
  Arms: eHealth Intervention

SUMMARY:
This trial will evaluate an eHealth breastfeeding co-parenting resource designed for mothers and their co-parents. Couples will be randomized to study groups and the intervention group will receive information about this resource or the control group will receive usual care. The primary outcomes will be exclusive breastfeeding at 4 and 24 weeks postpartum.

DETAILED DESCRIPTION:
This trial will evaluate an eHealth breastfeeding co-parenting resource designed for mothers and their co-parents. Couples will be randomized to study groups and the intervention group will receive information about this resource with an online demonstration and weekly emails for 6 weeks reminding them about the resource. The control group will receive usual care and 6 weekly emails reminding them that they are in the study. The primary outcomes will be exclusive breastfeeding at 4 and 24 weeks postpartum. Additional outcomes will include: breastfeeding initiation, duration, challenges, attitude, knowledge, confidence, anxiety, partners support and co-parenting.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, over 25 weeks pregnant, planning to breastfeed, lives with co-parent who is willing to participate, first time mother or mother who has not previously breastfed,

Exclusion Criteria:

* does not have access to the internet and telephone, does not reads and speaks English, does not lives in Ontario, Canada, is expecting more than one child with this pregnancy

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Infant Feeding Questionnaire | 4 weeks
  The primary outcome for this study is the rate of exclusive breastfeeding at 4 weeks postpartum. This is defined as no food or liquid other than breast milk (not even water) given to the infant and includes feeding expressed breast milk. However, under this definition of exclusive breastfeeding, undiluted drops or syrups consisting of vitamins, minerals supplements or medicines are included (Breastfeeding Committee for Canada, 2006; WHO, 2010). Exclusive breastfeeding will be determined by asking the mother what she has fed her baby in the last 7 days and what she usually feeds her baby. In this trial exclusive breastfeeding will be consistent with full breastfeeding described by Labbok and Krasovec (1990).

SECONDARY OUTCOMES:
Breastfeeding Knowledge | baseline, 2 weeks post intervention, 4 weeks postpartum
  This outcome will be assessed using a questionnaire designed for this study by a literature review and a group of breastfeeding experts including both professionals and lay individuals. The questionnaire included 32 items with scores ranging from 0-32. Each correct response was given a score of 1. Higher scores indicate greater breastfeeding knowledge.
Breastfeeding Attitude | baseline, 2 weeks post intervention, 4 weeks postpartum
  Iowa Infant Feeding Attitude Scale (IIFAS) measures attitude towards infant feeding methods. This scale consists of 17 items that cover various dimensions of infant feeding. The respondent indicate they agreed or disagreed with each statement, on a five point Likert scale that ranges from strongly agree (5) to strongly disagree (1). The items are worded so that about half are favourable of each feeding method. Items that favour formula feeding are then reverse scored. The items total score range from 17-85 and the lower scores reflect a preference for formula feeding whereas the higher scores reflect a preference for breastfeeding. (de la Mora, Russell, Dungy, Losch & Dusdieker, 1999).
Breastfeeding Self-efficacy | baseline, 2 weeks post intervention, 4 weeks postpartum
  To measure this variable the Breastfeeding Self-Efficacy Scale - Short Form (BSES-SF; Dennis, 2003) will used. This instrument has 14 items. The response format is on a Likert scale, ranging from 'not at all confident' (1) to 'very confident' (5) where items are summed to produce a total score, ranging from 14 to 70, with higher scores indicating greater breastfeeding self-efficacy. (Dennis, 2003)
Anxiety | baseline, 2 weeks post intervention, 4 weeks postpartum, 12 weeks
  Mothers and co-parent will complete an Anxiety screening scale (GAD-7). This is a 7 item scale to measure generalized anxiety. The response format is on a Likert scale ranging from "not at all" (0) to "nearly every day" (3) where items are summed to produce a total score, ranging from 0 to 21, with higher scores indicating higher levels of generalized anxiety. (Spitzer, Kroenke, Williams & Löwe, 2006)
Partner support for infant feeding | 4 and 12 weeks postpartum
  A version of the Postpartum Partner Support Scale (PPSS) adapted for infant feeding is 22-item self-report instrument being used to assess partner infant-feeding-specific perceptions of support. This scale was developed to assess functional elements of support: appraisal/emotional, informational, and instrumental. Two items were included to examine negative support from the partner. Items are rated on a 4-point scale to produce a summative score ranging from 22 to 88, with higher scores indicating higher levels of infant feeding-specific partner support. (Dennis, Brown & Brennenstuhl, 2017)
Co-parenting infant feeding scale | 4 and 12 weeks postpartum
  Mother will complete a co-parenting infant feeding scale. This 15-item self-report instrument being used to assess co-parent infant feeding behaviours. This scale was developed to assess functional elements of breastfeeding coparenting framework. Items are rated on a 4-point scale to produce a summative score ranging from 15 to 60, with higher scores indicating higher levels of coparenting infant feeding behaviours. (Abbass-Dick & Dennis, 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Abbass-Dick, Principal Investigator — Ms.
Locations (1):
- University of Ontario Institute of Technology, Oshawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbass-Dick J, Xie F, Koroluk J, Alcock Brillinger S, Huizinga J, Newport A, Goodman WM, Dennis CL. The Development and piloting of an eHealth breastfeeding resource targeting fathers and partners as co-parents. Midwifery. 2017 Jul;50:139-147. doi: 10.1016/j.midw.2017.04.004. Epub 2017 Apr 18. PMID 28448858
- [Background] Abbass-Dick J, Dennis CL. Breast-feeding Coparenting Framework: A New Framework to Improve Breast-feeding Duration and Exclusivity. Fam Community Health. 2017 Jan/Mar;40(1):28-31. doi: 10.1097/FCH.0000000000000137. PMID 27870751
- [Background] Dennis CL, Brown HK, Brennenstuhl S. The Postpartum Partner Support Scale: Development, psychometric assessment, and predictive validity in a Canadian prospective cohort. Midwifery. 2017 Nov;54:18-24. doi: 10.1016/j.midw.2017.07.018. Epub 2017 Jul 29. PMID 28780475
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Abbass-Dick J, Dennis CL. Maternal and paternal experiences and satisfaction with a co-parenting breastfeeding support intervention in Canada. Midwifery. 2018 Jan;56:135-141. doi: 10.1016/j.midw.2017.10.005. Epub 2017 Oct 18. PMID 29101865
- [Background] Abbass-Dick J, Stern SB, Nelson LE, Watson W, Dennis CL. Coparenting breastfeeding support and exclusive breastfeeding: a randomized controlled trial. Pediatrics. 2015 Jan;135(1):102-10. doi: 10.1542/peds.2014-1416. Epub 2014 Dec 1. PMID 25452653
- [Background] de la Mora, A., Russell, D. W., Dungy, C.I., Losch, M., & Dusdieker, L. (1999). The Iowa Infant Feeding Attitude Scale: Analysis of reliability and validity. Journal of Applied Social Psychology, 29, 2362-2380.
- [Background] Labbok M, Krasovec K. Toward consistency in breastfeeding definitions. Stud Fam Plann. 1990 Jul-Aug;21(4):226-30. PMID 2219227
- [Background] World Health Oraniazation. (2010). Indicators for Assessing Infant and Child Feeding Practices: part two measurement. Malta: WHO
- [Background] Breastfeeding Committee for Canada. (2006). Breastfeeding Definitions and Data Collection Periods.